CLINICAL TRIAL: NCT01830699
Title: Rilonacept (Arcalyst ®) in the Treatment of Subacromial Bursitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keesler Air Force Base Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FKE20120016H
Record Dates: First submitted 2013-04-06; First posted 2013-04-12 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Subacromial Bursitis
Keywords: Rilonacept; Subacromial Bursitis treatment; Corticosteroid Injection
MeSH Terms: interventions — rilonacept; Adrenal Cortex Hormones; Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rilonacept (Active Comparator): 160 mg of rilonacept will be injected in the subacromial bursa of participants in this arm.
  Interventions: Drug: Rilonacept
- Corticosteroid (Placebo Comparator): 80 mg (2 cc of 40 mg/mL) Kenalog intra-bursal once
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: Rilonacept — 160 mg intra-bursal once
  Other Names: Arcalyst
  Arms: Rilonacept
Drug: Corticosteroid — 2 cc (40 mg/mL) triamcinolone intra-bursal once
  Other Names: Triamcinolone (Kenalog)
  Arms: Corticosteroid

SUMMARY:
To date no trials have been performed looking at whether or not intra-bursal injection of an IL-1 antagonist provides pain relief similar to that of a corticosteroid injection. The subcutaneous injection of anakinra, an IL-1 receptor antagonist, in patients with shoulder pain due to rotator cuff tendonitis and subacromial bursitis was efficacious in relieving pain but this information was presented as a case series in a letter to the editor format, so the validity of these results would require additional testing [Omoigui S, et al. 2004]. Based mainly on the data from the intra-articular administration of anakinra, there have not been any adverse trends in outcomes or safety to suggest that intra-bursal injection of rilonacept will carry an increase risk of adverse events. The purpose of this trial is to compare the improvement in pain and function of patients with clinical symptoms and signs of subacromial bursitis of rilonacept vs. corticosteroid injection (standard of care).

DETAILED DESCRIPTION:
Background: Subacromial bursitis is an inflammatory condition which is typically triggered by altered rotator cuff mechanics. One of the mainstays of therapy is corticosteroid injection. Given the inflammatory nature of subacromial bursitis coupled with prominence of interleukin-1 (IL-1) beta on histopathologic assessment of resected subacromial bursa, targeted anti-IL-1 therapy would be an attractive alternative to corticosteroid injection.

Hypothesis: One intra-bursal injection of the IL-1 trap rilonacept (Arcalyst ®), currently FDA approved for the treatment of cryopyrin associated periodic syndrome (CAPS), is non-inferior to intra-bursal corticosteroid injection at 4 weeks post-procedure.

Methods: This study is a prospective trial lasting a total of 4 weeks. Patients with typical symptoms and signs of subacromial bursitis are randomized to either corticosteroid injection prepared in the usual fashion in clinic vs. injection of rilonacept. Prior to injection of either medication patients will complete a QuickDASH Questionnaire and provide a verbal pain score from 0 to 10. The Quick DASH Questionnaire and verbal pain score are then completed within 2 duty days of injection, 2 weeks after injection, and 4 weeks after injection by phone.

Primary Outcome: Primary outcome is improvement in QuickDASH. Secondary outcomes are improvement in the verbal pain score and monitoring for infection or other complications from rilonacept administration.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age or older and at a minimum have a recent history (more than 3 days worth) of shoulder pain with moderate to severe tenderness to palpation over the subacromial bursa.

Exclusion Criteria:

* Allergies to lidocaine, marcaine, or kenalog.
* Allergies to rilonacept
* Flare of active inflammatory arthritis (such as a flare of Rheumatoid Arthritis)
* Gout or Pseudogout attack of the shoulder with subacromial tenderness
* Active infection
* Actively receiving chemotherapy, radiation therapy, or anticipating surgery for neoplasia
* Active myocardial infarction
* Clinical and/or radiographic evidence of a fracture (clavicular, humeral, or other).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Carroll, MD, Principal Investigator — Keesler Medical Center
Locations (1):
- Keesler Medical Center, Keesler Air Force Base, Mississippi, United States

REFERENCES:
- [Derived] Carroll MB, Motley SA, Wohlford S, Ramsey BC. Rilonacept in the treatment of subacromial bursitis: A randomized, non-inferiority, unblinded study versus triamcinolone acetonide. Joint Bone Spine. 2015 Dec;82(6):446-50. doi: 10.1016/j.jbspin.2015.02.009. Epub 2015 Jul 13. PMID 26184525

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment was from March 2013 to December 2013. Subjects were recruited from the Internal Medicine (IM) or IM Subspecialties Clinic at a single academic community-size hospital.
Pre-assignment Details: Please refer to inclusion and exclusion criteria.
Groups:
- Triamcinolone (Kenalog): A mixture of lidocaine without epinephrine, bupivicaine, and 80 mg of triamcinolone acetonide will be injected in the subacromial bursa.
  Corticosteroid (Triamcinolone (Kenalog) )
Period: Overall Study
Arm/Group | Triamcinolone (Kenalog) | Rilonacept
Started | 13 | 20
Completed | 13 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Prior to starting the trial, we anticipated having to recruit 150 subjects total (75 in each arm). At our first analysis of the data, the effect size of both the rilonacept and triamcinolone were larger than expected, and a re-calculated 'n' was 29 for an alpha of 0.05 and power of 1.0000 (effect size 1.1).
Groups:
- Total: Total of all reporting groups
Arm/Group | Triamcinolone (Kenalog) | Rilonacept | Total
Number analyzed (Participants) | 13 | 20 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (13.7) | 64.5 (12.1) | 65.3 (12.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 12 | 18
  >=65 years | 7 | 8 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 11 | 19 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 20 | 33
Site of subacromial injection [Number; unit: participants]
  Right Bursa injected | 6 | 14 | 20
  Left Bursa injected | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Shoulder Function
Description: The QuickDASH will be used as the primary outcome to assess improvement in pain and function of patients with clinical symptoms and signs of subacromial bursitis randomized to either rilonacept vs. corticosteroid injection. The QuickDASH is an 11 question form, a short version of the Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH). It ranges from 0 (no symptoms/full function) to 100 (maximal symptoms/no function). No units are specified. Cutoff scores: < 15 = no problem, 16 - 40 = problem, but working, > 40 = unable to work. US population mean +/- SD is 10.1 +/- 14.7.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triamcinolone (Kenalog) | Rilonacept
Number analyzed (Participants) | 13 | 20
units on a scale | 15.92 (15.40) | 38.52 (25.07)
Statistical Analysis 1: Comparison: Triamcinolone (Kenalog) vs Rilonacept; Setting α=0.05 and β=0.8, with effect size of 0.17 anticipated total n = 138 to be recruited (requested recruitment of 150 to account for possible drop-outs) 1st data analysis (n = 33), effect size calculated at 1.1 with new n = 29 with α=0.05 and β=1.0; Test type: Non-Inferiority or Equivalence — For details of power calculation, see above. Using a minimal clinical importance of -9.1, the null hypothesis was a mean difference less than -9.1; p = 0.004, t-test, 2 sided; Mean Difference (Final Values) = -23.9

2. Secondary Outcome: Improvement in Pain
Description: Secondary outcomes are improvement in pain (as assessed by patient self report, range between 0 and 10, with 0 as no pain and 10 described as the worst pain in their life).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triamcinolone (Kenalog) | Rilonacept
Number analyzed (Participants) | 13 | 20
units on a scale | 2.27 (1.42) | 3.85 (2.74)
Statistical Analysis 1: Comparison: Triamcinolone (Kenalog) vs Rilonacept; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — See details above regarding effect size, power, etc; p = 0.044, t-test, 2 sided

3. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Any adverse event reported by the study participant during the four time points studied in the trial in either arm will be recorded.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Triamcinolone (Kenalog) | Rilonacept
Number analyzed (Participants) | 13 | 20
participants | 3 | 8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Triamcinolone (Kenalog) | Rilonacept
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/20
Other Adverse Events (participants affected / at risk) | 2/13 | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triamcinolone (Kenalog) (N=12) | Rilonacept (N=20)
Hospitalization (Infections and infestations) | 1 (12) | 1 (20) — One subject in the rilonacept arm was hospitalized for diarrhea, heme-occult positive stool, and an INR of 3.4. One subject in the triamcinolone arm was hospitalized for shortness of breath for which an etiology was never identified.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triamcinolone (Kenalog) (N=13) | Rilonacept (N=20)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Injection Site Reaction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Acute Bronchitis (Infections and infestations) | 0 (0) | 1 (1) — Required antibiotics
Generalized Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hand Tingling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes